CLINICAL TRIAL: NCT01763606
Title: A Pilot Trial of Enoxaparin Versus Aspirin in Patients With Cancer and Stroke
Brief Title: Enoxaparin Versus Aspirin in Patients With Cancer and Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Presbyterian Hospital (Other); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-264
Record Dates: First submitted 2012-12-20; First posted 2013-01-09 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2019-04

CONDITIONS: Cancer Patients First-ever Acute Ischemic Stroke
Keywords: Enoxaparin; Aspirin; stroke; 12-264
MeSH Terms: conditions — Stroke | interventions — Enoxaparin; Aspirin

ARMS (2):
- Enoxaparin (Experimental): Patients assigned to enoxaparin.
  Interventions: Drug: Enoxaparin
- Aspirin (Experimental): Patients assigned to Aspirin.
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Enoxaparin — Patients will be receive 6 months of subcutaneous enoxaparin (1 mg/kg BID with a maximum starting dose of 100 mg BID. Patients who weigh more than 100 kg will start at a dose of 100 mg BID; their subsequent dosing will be guided by hematology and may change.
  Arms: Enoxaparin
Drug: Aspirin — Patients will receive 6 months of oral aspirin (81 mg per day unless a higher dose is preferred by study physicians although the maximum acceptable dose will be 325 mg per day).
  Arms: Aspirin

SUMMARY:
Patients with cancer who develop stroke are at high risk for future strokes or other clotting events. These patients are routinely treated with medicines that thin their blood, including enoxaparin or aspirin. However, it is unclear which medicine is best and whether these medicines can be adequately studied in a clinical trial.

The purpose of this Phase I/II study is to determine if a clinical trial of different blood thinners in patients with cancer and stroke is possible. In addition, the study aims to compare the effects, good and/or bad, of enoxaparin with those of aspirin on patients with cancer and recent stroke.

ELIGIBILITY:
Any adult patient with active systemic cancer diagnosed with acute ischemic stroke at the main MSKCC campus or at any of MSKCC's New York City outpatient center WCMC, NYPH/CUMC within the prior four weeks would be eligible.

Inclusion Criteria:

* 18 to 85 years of age.
* Active cancer, defined as a pathologic diagnosis of or treatment for any cancer, other than basal-cell or squamous-cell carcinoma of the skin, within the past six months; or patients with known recurrent or metastatic disease within the past six months.
* A pathology report issued at the enrolling site confirming the diagnosis of cancer is required for enrollment.
* Acute ischemic stroke within the prior four weeks, defined as a new neurologic deficit(s) with MRI evidence of acute ischemia in a referable location, and no clinical or radiologic indication of a non-cerebrovascular mimic, such as a brain metastasis, as the etiology of the deficit(s).

Exclusion Criteria:

* Inability to get brain MRI
* Known malignant primary brain tumor.
* Diagnosis of intracranial hemorrhage within the past 3 months, including intratumoral hemorrhage into brain metastases from a systemic cancer.
* Active or serious bleeding within two weeks of enrollment.
* Patient condition associated with a high risk of bleeding such as recent surgery or peptic ulcer disease.
* Clear indication for anticoagulation (e.g., atrial fibrillation) anticipated during the study period.
* Clear indication for antiplatelet agents (e.g., cardiac stents); a patient receiving aspirin for primary prevention prior to index stroke may be enrolled as long as study investigators believe it would be safe for the patient to stop aspirin if the patient was randomized to the enoxaparin arm.
* Active bleeding diathesis.
* Platelet count of ≤ 70,000/mm3, an international normalized ratio (INR) > 1.6, or a partial thromboplastin time (PTT) > 40 seconds.
* Known allergy to heparin or aspirin or a history of heparin induced thrombocytopenia.
* Serum creatinine > 2 mg/dl.
* AST or ALT > 200 U/L.
* Hemoglobin < 8 gm/dl
* Symptomatic carotid stenosis.
* Active pregnancy.
* Life expectancy < 1 month or current hospice care
* Unavailability for follow-up.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-12-18 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2019-04-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa DeAngelis, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering West Harrison, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Columbia University, New York, New York
  - Weill Cornell Medical Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Enoxaparin | Aspirin
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enoxaparin | Aspirin | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Full Range); unit: years] | 68 [54 to 75] | 71 [63 to 81] | 71 [54 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 10 | 20
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 4 | 8 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Safety Outcomes
Description: Number of Participants with intracranial hemorrhage, symptomatic intracranial hemorrhage, major bleeding, and death
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin | Aspirin
Number analyzed (Participants) | 10 | 10
Participants
  Fatal Recurrent AIS | 1 | 0
  Nonfatal gastrointestinal bleeding | 0 | 3
  Nonfatal pulmonary hemorrhage | 1 | 0
  No hemorrahage, major bleeding or death | 8 | 7

2. Primary Outcome: Feasibility Outcomes
Description: The primary feasibility outcome is patient enrollment defined as the number of patients who enroll in the study divided by the number of patients who were eligible to enroll.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: percentage of eligible pts enrolled
Groups:
- Eligible Participants: Participants eligible for study
Arm/Group | Eligible Participants
Number analyzed (Participants) | 49
percentage of eligible pts enrolled | 41 [27 to 55]

3. Secondary Outcome: Number of Participants With or Without Recurrent Ischemic Stroke
Description: Secondary efficacy outcomes will be assessed for and will include recurrent ischemic stroke, all strokes (ischemic or hemorrhagic), transient ischemic attack, myocardial infarction, deep vein thrombosis, pulmonary embolism, and systemic arterial thrombosis. Functional outcomes will also be evaluated, including the modified Rankin Scale score, the National Institute of Health Stroke Scale, and the Karnofsky Performance Status Scale.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Enoxaparin | Aspirin
Number analyzed (Participants) | 10 | 10
Participants
  Recurrent ischemic event | 1 | 0
  No recurrent ischemic event | 9 | 10

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Enoxaparin | Aspirin
All-Cause Mortality (participants affected / at risk) | 6/10 | 6/10
Serious Adverse Events (participants affected / at risk) | 5/10 | 6/10
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enoxaparin (N=10) | Aspirin (N=10)
Constipation (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 1
Death NOS (General disorders) | 0 | 2
Dysphasia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enoxaparin (N=10) | Aspirin (N=10)
Alanine aminotransferase increased (Investigations) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 2
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Stroke (Nervous system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
White blood cell decreased (Investigations) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 2
Confusion (Psychiatric disorders) | 0 | 1
Dysphasia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-06): https://cdn.clinicaltrials.gov/large-docs/06/NCT01763606/Prot_SAP_000.pdf